CLINICAL TRIAL: NCT05436249
Title: Using Motor Imagery and Machine Learning-Based Real-Time fMRI Neurofeedback to Improve Motor Function in Cerebellar Ataxia
Brief Title: Use of Real-Time Functional Magnetic Resonance Imaging Neurofeedback to Improve Motor Function in Cerebellar Ataxia
Acronym: fMRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other); Johns Hopkins Discovery Award (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: IRB00281329
Record Dates: First submitted 2022-06-23; First posted 2022-06-29 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Cerebellar Ataxia; Healthy Controls; Ataxia; Spinocerebellar Ataxias; Cerebellar Diseases; Neurodegenerative Diseases; Movement Disorders; Cerebellum; Gait; Balance
MeSH Terms: conditions — Cerebellar Ataxia; Ataxia; Spinocerebellar Ataxias; Cerebellar Diseases; Neurodegenerative Diseases; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real time neurofeedback with task (Other): Participants will undergo a real-time fMRI scan during which two distinct tasks will be performed.
  Interventions: Device: Neurofeedback treatment
- Overt tapping and/or motor imagery practice (Other): Participants will undergo an overt tapping task at baseline. Participants are assigned to a group where they will then perform respective motor and/or imagery tasks at home for 3 weeks.
  Interventions: Behavioral: At-home therapy

INTERVENTIONS:
Device: Neurofeedback treatment — During the fMRI scan, the tasks consist of:
  1. Overt finger tapping in time with a flashing cue.
  2. Motor imagery (of finger tapping).
  During overt finger tapping, feedback will consist of a slider bar that indicates tapping accuracy to target speed (1 or 4Hz). During motor imagery, neurofeedback will consist of a slider bar that indicates the success of recruiting predicted brain regions (consistent with those engaged during overt tapping).
  Arms: Real time neurofeedback with task
Behavioral: At-home therapy — Participants are assigned to groups where they will practice each day for 3 weeks at-home.
  1. Group 1: Imagery only.
  2. Group 2: Overt finger tapping only.
  3. Group 3: Imagery plus overt finger tapping.
  During imagery, participants will view the task while imagining that they are finger tapping in time with the flashing cue, using the imagery strategies identified during their previous neurofeedback session. During overt tapping, participants will finger tap in time with the flashing cue. A final assessment of overt tapping will be performed the day after therapy ends.
  Arms: Overt tapping and/or motor imagery practice

SUMMARY:
This project will study the feasibility of motor rehabilitation in people with cerebellar ataxia using real-time functional magnetic resonance imaging neurofeedback (rt-fMRI NF) in conjunction with motor imagery. To do so, data will be collected from healthy adults in this protocol, to be compared with data from cerebellar ataxia participants.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years of age
* At least 8th-grade education
* Right-handedness

Exclusion Criteria:

* History of Axis I psychiatric disorders (including alcohol and drug dependence)
* Severe or unstable medical disorder, neurological disorders, such as stroke or epilepsy
* History of head injury that resulted in a loss of consciousness greater than 5 minutes and/or neurological sequelae
* Any condition that is contraindicated for the MRI environment (e.g., metal in the body, pacemaker, claustrophobia)
* Currently pregnant
* Eligible subjects may be asked to refrain from medications that affect the central nervous system that would also make data difficult to interpret (e.g., sedatives) for an appropriate period of time prior to scanning
* Participants will be excluded if they do not have a home computer with internet available to complete the 3-week at-home component of the study protocol

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2023-12-28 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Change in overt tapping accuracy as assessed by finger tapping to a flashing cue at 1Hz speed | Baseline and MRI duration, up to 1 hour
  During the MRI session, accuracy on overt tapping will be measured by the distance of the actual tapping rate vs. target rate (1Hz). Accuracy at baseline will be compared to that of final assessment, which will take place before and after neurofeedback training, respectively. The difference in accuracy between the two tests create a delta measure (i.e., fewer errors in the final vs. baseline tests). This delta accuracy will indicate the magnitude of tapping accuracy improvements. Root mean squared error (RMSE) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 1 tap for 1Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Change in overt tapping accuracy as assessed by finger tapping to a flashing cue at 4Hz speed | Baseline and MRI duration, up to 1 hour
  During the MRI session, accuracy on overt tapping will be measured by the distance of the actual tapping rate vs. target rate (4Hz). Accuracy at baseline will be compared to that of final assessment, which will take place before and after neurofeedback training, respectively. The difference in accuracy between the two tests create a delta measure (i.e., fewer errors in the final vs. baseline tests). This delta accuracy will indicate the magnitude of tapping accuracy improvements. RMSE (root mean squared error) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 4 taps for 4Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Change in at-home overt tapping accuracy as assessed by finger tapping to a flashing cue at 1Hz speed | Baseline and At-home sessions (10 minutes/day), up to 23 days
  Accuracy at baseline will be compared to that of final assessment, which will take place before and after the 3-week at-home practice sessions, respectively. The delta measure will indicate the magnitude of tapping accuracy improvements. Groups will be compared to examine differences in delta as a function of practice condition (imagery only, tapping only, or imagery plus tapping). At-home tapping performance will be compared to MRI tapping performance. RMSE (root mean squared error) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 1 tap for 1Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.
Change in at-home overt tapping accuracy as assessed by finger tapping to a flashing cue at 4Hz speed | Baseline and At-home sessions (10 minutes/day), up to 23 days
  Accuracy at baseline will be compared to that of final assessment, which will take place before and after the 3-week at-home practice sessions, respectively. The delta measure will indicate the magnitude of tapping accuracy improvements. Groups will be compared to examine differences in delta as a function of practice condition (imagery only, tapping only, or imagery plus tapping). At-home tapping performance will be compared to MRI tapping performance. RMSE (root mean squared error) is the measure for both the baseline and post-treatment behavioral tasks. RMSE will be based on the actual number of taps per second relative to the expected number of taps per second (e.g., 4 taps for 4Hz). Then post treatment RMSE minus baseline RMSE will determine a delta RMSE. A higher RMSE signifies greater error. For the delta measure, it is expected, lower scores reflect greater improvement on the task.

SECONDARY OUTCOMES:
The correlation between MRI BOLD and finger tapping accuracy to a flashing cue at 1Hz as assessed by a correlation coefficient | MRI duration, up to 1 hour
  This will assess the correlation between MRI Blood Oxygen Level Dependence (BOLD) and finger tapping accuracy by a correlation coefficient. The correlation coefficient ranges from -1 to 1, where the closer the coefficient is to -1 indicates a strong negative association and the closer the coefficient is to 1 indicates a strong positive association.
The correlation between MRI BOLD and finger tapping accuracy to a flashing cue at 4Hz as assessed by a correlation coefficient | MRI duration, up to 1 hour
  This will assess the correlation between MRI BOLD (Blood Oxygen Level Dependence) and finger tapping accuracy by a correlation coefficient. The correlation coefficient ranging from -1 to 1, where the closer the coefficient is to -1 indicates a negative association and the closer the coefficient is to 1 indicates a strong positive association.
The correlation between the KVIQ and imagery accuracy of the slider bar from target on the MRI task as assessed by a correlation coefficient | Up to 1.5 hours
  The Kinesthetic and Visual Imagery Questionnaire (KVIQ), overall score ranging from 0-100, where higher scores reflect more vivid imagery) will assess imagery vividness. This will be correlated with the image accuracy measures described in Secondary Outcome Measure 5'.
The correlation between the ICARS and imagery accuracy of the slider bar from target on the MRI task as assessed by a correlation coefficient | Up to 1.5 hours
  The International Cooperative Ataxia Rating Scale (ICARS), overall score ranging from 0-100, where higher scores indicate more severe neurological impairment) will assess neurological impairments. This will be correlated with image accuracy measures described in 'Secondary Outcome Measure 5'.

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Marvel, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Immediately following publication. No end date.
Access Criteria: Access to trial individual participant data (IPD) can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact cmarvel1@jhmi.edu.